CLINICAL TRIAL: NCT00485173
Title: A Pivotal Clinical Investigation of INFUSE® Bone Graft With a PEEK Interbody Spacer and an Anterior Cervical Plate in Patients With Cervical Degenerative Disc Disease at a Single Level.
Brief Title: INFUSE® Bone Graft/ PEEK Interbody Spacer/ Anterior Cervical Plate Pivotal Clinical Trial
Acronym: ACDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFUSE® Bone Graft PEEK ACDF
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2012-12

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- INFUSE® Bone Graft (Experimental): In this arm, patients will receive implant with INFUSE® Bone Graft/PEEK Spacer/Anterior Cervical Plate.
  Interventions: Device: INFUSE® Bone Graft/PEEK Spacer/Anterior Cervical Plate

INTERVENTIONS:
Device: INFUSE® Bone Graft/PEEK Spacer/Anterior Cervical Plate — All patients enrolled in this study will receive the investigational device.
  Other Names: ACDF, Anterior Cervical Plate

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the investigational implant (INFUSE® Bone Graft/PEEK Interbody Spacer/Anterior Cervical Plate) as a method of facilitating spinal fusion at a single level from C3-C7 in patients with symptomatic cervical degenerative disc disease.

DETAILED DESCRIPTION:
This pivotal clinical trial is being conducted to evaluate the safety and effectiveness of INFUSE® Bone Graft with the PEEK Interbody Spacer and Anterior Cervical Plate in patients with symptomatic cervical degenerative disc disease (DDD). The implant under investigation in this clinical trial is INFUSE® Bone Graft, the PEEK Interbody Spacer, and Anterior Cervical Plate. The device will be implanted using an anterior surgical approach. Safety and effectiveness data for patients in this study will be compared to that of historical controls. Historical control data will be taken from the control arms of the following Medtronic studies: (1) the Artificial Cervical Disc (also known as PRESTIGE® Cervical Disc System) pivotal IDE trial (NCT00642876) and (2) the BRYAN® Cervical Disc System pivotal IDE trial (NCT00437190).

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION:

  1. Single-level cervical degenerative disc disease (from C3-C7) requiring surgical treatment and involving intractable radiculopathy and/or myelopathy.
  2. Herniated disc and/or osteophyte formation at the level to be treated that is producing symptomatic nerve root and/or spinal cord compression.
  3. Unresponsive to non-operative treatment for six weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management.
  4. At least 18 years of age and skeletally mature at the time of surgery.
  5. A preoperative Neck Disability Index (NDI) score ≥30.
  6. A preoperative neck pain score (pain intensity + pain frequency) ≥8 (out of 20) based on the preoperative Neck and Arm Pain Questionnaire.
  7. If a female of childbearing potential, patient is not pregnant or nursing and agrees not to become pregnant for one year following surgery.
  8. Is willing and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* EXCLUSION:

  1. A cervical spinal condition other than symptomatic cervical degenerative disc disease requiring surgical treatment at the involved level.
  2. Documented or diagnosed cervical instability at the target level, defined by dynamic (flexion/extension) radiographs.
  3. Previous surgical intervention at the involved level.
  4. Any subsequent planned/staged surgical procedure at the involved or adjacent level(s).
  5. Fused level adjacent to the level to be treated.
  6. Severe pathology of the facet joints of the involved vertebral bodies.
  7. Has osteoporosis, osteopenia, or osteomalacia as determined by DEXA scan.
  8. Presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
  9. Overt or active bacterial infection, either local or systemic.
  10. Insulin dependent diabetes.
  11. Chronic or acute renal failure or prior history of renal disease.
  12. Documented allergy or intolerance to stainless steel, titanium, titanium alloy, polyetheretherketone (PEEK), or tantalum.
  13. Is mentally incompetent. (if questionable, obtain psychiatric consult.)
  14. Is a prisoner.
  15. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
  16. On oral or injectable steroids for 6 weeks or more at the time of enrollment.
  17. A history of autoimmune disease.
  18. History of exposure to injectable collagen or silicone implants.
  19. History of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
  20. Received any previous exposure to any/all BMPs either human or animal extraction.
  21. History of allergy to bovine products.
  22. History of any allergy resulting in anaphylaxis.
  23. History of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers-Danlos Syndrome, or osteogenesis imperfecta).
  24. Condition that requires postoperative medications that interfere with the stability of the implant, such as steroids.
  25. Received treatment with an investigational therapy (drug, device, or biologic) within 28 days prior to implantation surgery or such treatment is planned during the 24-month period following the study surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - S & B Surgery Center, Beverly Hills, California
  - Orange County Neurological Association, Laguna Hills, California
  - Crane Creek Medical Ctr. The Back Center /Osler Medical, Melbourne, Florida
  - The Hughston Clinic, P.C., Columbus, Georgia
  - University of Kansas Medcal Center, Kansas City, Kansas
  - Spine Institute, Shreveport, Louisiana
  - Springfield Neurological Institute, Springfield, Missouri
  - Buffalo Neurosurgery Group, West Seneca, New York
  - University of Cincinnati Dept of Neurosurgery, Cincinnati, Ohio
  - TriState Orthopedic Treatment Center, Norwood, Ohio
  - The Washington Hospital, Washington, Pennsylvania
  - Center for Sports Medcine & Orthopedics, Chattanooga, Tennessee
  - Semmes Murphey Neurologic & Spine Institute, Memphis, Tennessee
  - Central Texas Spine, Austin, Texas
  - Brain and Spine Center of Texas, L.L.P., Plano, Texas
  - Inland Neurosurgery & Spine Associates, P.S., Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five subjects in investigational group and 4 subjects in control group died within 24 months postoperatively. Among them, however, one investigational subject who died at 20 months and one control subject who died at 23 months reported some data that were included as the 24-month evaluation. Thus, they were counted as evaluated at 24 months.
Groups:
- INFUSE® Bone Graft: In this arm, patients received implant with INFUSE® Bone Graft/PEEK Spacer/Anterior Cervical Plate.
- Historical Control: Historical control was pooled from the control arms of the following Medtronic studies: (1) the Artificial Cervical Disc (also known as PRESTIGE® Cervical Disc System) pivotal IDE trial (NCT00642876) and (2) the BRYAN® Cervical Disc System pivotal IDE trial (NCT00437190).
Period: Overall Study
Arm/Group | INFUSE® Bone Graft | Historical Control
Started | 224 | 486
Completed | 188 (The number of completed participants is reported the number of subjects who had any 24-month data.) | 422 (The number of completed participants is reported the number of subjects who had any 24-month data.)
Not Completed | 36 | 64
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 32 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INFUSE® Bone Graft | Historical Control | Total
Number analyzed (Participants) | 224 | 486 | 710
Age Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.2) | 44.2 (8.7) | 45.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 251 | 369
  Male | 106 | 235 | 341
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 198 | 447 | 645
  Black | 20 | 18 | 38
  Asian | 2 | 4 | 6
  Hispanic | 3 | 13 | 16
  Other | 1 | 4 | 5
Height [Mean (Standard Deviation); unit: in.] | 67.5 (4.2) | 67.5 (4.0) | 67.5 (4.1)
Weight [Mean (Standard Deviation); unit: lbs.] | 188.8 (43.6) | 182.5 (40.4) | 184.5 (41.5)
Marital Status [Number; unit: participants]
  Single | 30 | 61 | 91
  Married | 163 | 373 | 536
  Divorced | 21 | 44 | 65
  Separated | 7 | 4 | 11
  Widowed | 3 | 4 | 7
Education Level [Number; unit: participants]
  < high School | 10 | 29 | 39
  High School | 80 | 142 | 222
  > high School | 134 | 314 | 448
Worker's Compensation [Number; unit: participants]
  Yes | 5 | 46 | 51
  No | 219 | 440 | 659
Unresolved Spinal Litigation [Number; unit: participants]
  Yes | 28 | 38 | 66
  No | 196 | 448 | 644
Tobacco Used [Number; unit: participants]
  Yes | 66 | 145 | 211
  No | 157 | 341 | 498
Alcohol Used [Number; unit: participants]
  Yes | 111 | 150 | 261
  No | 113 | 336 | 449
Preop Work Status [Number; unit: participants]
  Yes | 153 | 309 | 462
  No | 71 | 176 | 247

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Success
Description: Rate of overall success is reported as the percentage of participants who met all of the following criteria:
  1. fusion at the treated level;
  2. pain/disability (Neck Disability Index) success;
  3. neurological status success;
  4. no serious adverse event classified as "implant associated" or "implant/surgical procedure associated;"
  5. no additional surgical procedure classified as a "failure."
Time Frame: 24 months post-operation
Population: Primary dataset (including all subjects who received study devices. Missing observations were not imputed.)
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 162 | 352
percentage of participants | 80.9 | 59.9
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — P-value was one-sided from random samplings, based on logistic regression model by using propensity score as a covariate
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority comparison of success rates in two treatment groups was a secondary objective of this trial. Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

2. Secondary Outcome: Success Rate of Fusion
Description: Success Rate of Fusion is reported as percent of participants who met the following fusion criteria:
  1. Evidence of bridging bone. This is based on the evidence of a continuous bony connection from the superior vertebral body to the inferior vertebral body in at least one of the following areas: lateral, anterior, posterior and/or through the PEEK spacer.
  2. No evidence of radiolucency at greater than 50% of the superior or inferior PEEK spacer-vertebra interface.
  3. No evidence of motion as defined by ≤ 4º of angular motion (based on flexion-extension lateral plain radiographs).
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 160 | 345
percentage of participants | 99.4 | 87.2
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.002, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

3. Other Pre Specified Outcome: Neck Disability Index Score
Description: The self-administered Neck Disability Index (NDI) Questionnaire was used to assess patient neck pain and ability to function. The NDI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 413
units on a scale
  NDI at baseline | 50.2 (14.3) | 53.5 (16.2)
  NDI at 24 months | 14.6 (17.1) | 20.9 (16.0)
  NDI change at 24 months from baseline | -34.9 (17.3) | -32.3 (20.9)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was one-sided, adjusted from ANCOVA with the propensity score as the covariate

4. Secondary Outcome: Success Rate of Neck Disability Index
Description: Success rate of Neck Disability Index is reported as the percentage of participants whose neck disability index score met: Pre-treatment Score - Post-treatment Score ≥ 15.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 413
percentage of participants | 85.8 | 79.9
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — P-value was one-sided from random sampling, based on covariance matrix produced by logistic regression using propensity score as a covariate
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.011, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

5. Other Pre Specified Outcome: Neck Pain Score
Description: Numerical rating scales are used to evaluate neck pain intensity and frequency. Patients rate their neck pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients record their neck pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total neck pain score is the sum of pain intensity and frequency scores.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 175 | 413
units on a scale
  Neck pain at baseline | 15.9 (2.7) | 15.8 (3.8)
  Neck pain at 24 months | 4.5 (5.2) | 6.0 (6.9)
  Neck pain change at 24 months from baseline | -11.2 (5.3) | -9.8 (7.2)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.063, ANCOVA — P-value was one-sided, adjusted from ANCOVA with the propensity score as the covariate

6. Secondary Outcome: Success Rate of Neurological Status
Description: Success rate of neurological status is reported as the percentage of participants who met neurological success defined as maintenance or improvement in all sections (motor, sensory, and reflexes) for the time period evaluated. In order for a section to be considered a success, each element in the section must remain the same or improve from the time of the preoperative evaluation to the time period evaluated.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 177 | 414
percentage of participants | 93.8 | 85.0
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

7. Other Pre Specified Outcome: Arm Pain Score
Description: Numerical rating scales are used to evaluate arm pain intensity and frequency. Patients rate their arm pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients record their arm pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total arm pain score will be the sum of pain intensity and frequency scores.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 175 | 413
units on a scale
  Arm pain at baseline | 13.5 (5.1) | 14.8 (4.7)
  Arm pain at 24 months | 3.6 (4.9) | 4.7 (5.8)
  Arm pain change at 24 months from baseline | -10.1 (6.3) | -10.1 (6.9)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value was one-sided, adjusted from ANCOVA with the propensity score as the covariate

8. Secondary Outcome: Neck Pain Success Rate
Description: Neck pain success rate is reported as the percentage of participants whose neck pain improvement met: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 175 | 413
percentage of participants | 96.0 | 92.7
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p = 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.414, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

9. Other Pre Specified Outcome: General Health Status -- SF-36 PCS
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results are summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 407
units on a scale
  SF-36 PCS at baseline | 31.6 (6.6) | 31.9 (7.3)
  SF-36 PCS at 24 months | 47.7 (11.1) | 45.3 (11.5)
  SF-36 PCS change at 24 months from baseline | 15.6 (10.9) | 13.1 (11.2)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value was one-sided, adjusted from ANCOVA with the propensity score as the covariate

10. Secondary Outcome: Arm Pain Success Rate
Description: Arm pain success rate is reported as the percentage of participants whose arm pain improvement met: Preoperative Score - Postoperative Score > 0.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 175 | 413
percentage of participants | 90.9 | 88.6
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.017, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

11. Other Pre Specified Outcome: General Health Status -- SF-36 MCS
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results are summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for MCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 407
units on a scale
  SF-36 MCS at baseline | 43.6 (12.0) | 43.6 (12.1)
  SF-36 MCS at 24 months | 51.8 (9.5) | 50.9 (10.8)
  SF-36 MCS Change at 24 months from baseline | 8.0 (12.0) | 7.2 (13.4)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.189, ANCOVA — P-value was one-sided, adjusted from ANCOVA with the propensity score as the covariate

12. Secondary Outcome: Success Rate of SF-36 PCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success rate of SF-36 PCS was defined as: Post Score - Pre Score >= 0.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 407
percentage of participants | 89.8 | 88.2
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.466, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

13. Secondary Outcome: Success Rate of SF-36 MCS
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success rates of SF-36 MCS were defined as: Post Score - Pre Score >= 0.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 176 | 407
percentage of participants | 75.0 | 71.3
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.10; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: INFUSE® Bone Graft vs Historical Control; Superiority analysis was performed if non-inferiority was demonstrated; Test type: Superiority or Other; p = 0.133, Regression, Logistic — P-value was one-sided, obtained from logistic regression model by using propensity score as a covariate

14. Secondary Outcome: Operative Time
Description: Operative time was recorded from skin incision to wound closure.
Time Frame: Time of operation, approximately 1.5 hrs.
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 224 | 486
hrs | 1.0 (0.5) | 1.4 (0.6)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was two-sided, adjusted from ANCOVA with the propensity score as the covariate

15. Secondary Outcome: Blood Loss
Time Frame: During the time of operation, approximately 1.5 hours.
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 224 | 484
ml | 40.1 (54.1) | 58.4 (59.9)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was two-sided, adjusted from ANCOVA with the propensity score as the covariate

16. Secondary Outcome: Hospital Stay
Time Frame: During the time of hospital stay, average of 1 day.
Population: Primary dataset.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 224 | 486
days | 1.0 (0.7) | 1.0 (0.6)
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.341, ANCOVA — P-value was two-sided, adjusted from ANCOVA with the propensity score as the covariate

17. Secondary Outcome: Number of Patients Who Had Secondary Surgeries at the Index Level
Description: Secondary surgical procedures at the index level included revisions, removal, supplemental fixation and reoperations.
Time Frame: 24 months post-operation
Measure: Number; unit: participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 224 | 486
participants | 6 | 27
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Test type: Superiority or Other; p = 0.479, Regression, Cox — P-value was two-sided, obtained from Cox regression and adjusted with propensity scores

18. Other Pre Specified Outcome: Ossification in the Region of Target Level
Description: Ossification in the region of target level is reported as the percentage of the patients who had ossification in the region of the target level. The region of target level included the index level, the superior and inferior adjacent disc spaces, and the superior and inferior adjacent vertebral bodies.
Time Frame: 24 months post-operation
Population: Primary dataset.
Measure: Number; unit: percentage of participants
Arm/Group | INFUSE® Bone Graft | Historical Control
Number analyzed (Participants) | 224 | 486
percentage of participants
  Preoperative (n=220, 442) | 40.9 | 36.9
  24 months (n=168, 407) | 78.6 | 59.2
Statistical Analysis 1: Comparison: INFUSE® Bone Graft vs Historical Control; Statistical analysis at 24 months postoperation; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value was from logistic regression model by using propensity score and any ossification 'Yes/No' at preop as the covariates

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | INFUSE® Bone Graft | Historical Control
Serious Adverse Events (participants affected / at risk) | 71/224 | 159/486
Other Adverse Events (participants affected / at risk) | 186/224 | 371/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE® Bone Graft (N=224) | Historical Control (N=486)
Acute Myoccardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid Cyst (Endocrine disorders) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Ectropion (Eye disorders) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Accidental Death (General disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Axillary Pain (General disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 3 (3)
Device Breakage (General disorders) | 0 (0) | 1 (1)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 3 (3) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Soft Tissue Inflammation (General disorders) | 1 (1) | 0 (0)
Spinal Pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Immunodeficiency Common Variable (Immune system disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Extradural Abscess (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Herpes (Infections and infestations) | 0 (0) | 1 (1)
Paraoesophageal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Primary Atypical (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Accident At Work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone Fragmentation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epidural Fibrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 6 (6)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral Disc Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus Lesion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Multiple Drug Overdose Accidental (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal Deviation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1)
Pancreatic Enzymes Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 15 (15)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 12 (16)
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 9 (9) | 18 (18)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 15 (15) | 32 (35)
Intervertebral Disc Space Narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ligament Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (10)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 16 (18)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 16 (16)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 5 (6) | 11 (12)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoid Cyst (Nervous system disorders) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 2 (2) | 10 (10)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 7 (7)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dysaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 8 (9)
Hypokinesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 3 (3) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Myelitis Transverse (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Nerve Root Compression (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (4)
Perineurial Cyst (Nervous system disorders) | 1 (1) | 1 (1)
Radicular Pain (Nervous system disorders) | 0 (0) | 7 (7)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sensory Loss (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 1 (1) | 3 (3)
Spinal Cord Ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Oedema (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Thoracic Outlet Syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Ulnar Nerve Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Foetal Hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus Ureteric (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis Interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Neurogenic Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular Torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Foreign Body Aspiration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal Haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Keloid Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Face Lift (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE® Bone Graft (N=224) | Historical Control (N=486)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 5 (5)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 3 (3) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1) | 2 (2)
Vitreous Floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breath Odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Change Of Bowel Habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 34 (37) | 34 (36)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (4) | 7 (7)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malocclusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 8 (8)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Polyp Colorectal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue Discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5)
Adverse Drug Reaction (General disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 5 (6) | 0 (0)
Axillary Pain (General disorders) | 0 (0) | 2 (2)
Chest Discomfort (General disorders) | 0 (0) | 2 (2)
Chest Pain (General disorders) | 2 (2) | 10 (10)
Chills (General disorders) | 1 (1) | 0 (0)
Crepitations (General disorders) | 1 (1) | 1 (1)
Device Breakage (General disorders) | 0 (0) | 3 (3)
Device Connection Issue (General disorders) | 0 (0) | 2 (2)
Device Dislocation (General disorders) | 0 (0) | 1 (1)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 1 (1)
Feeling Cold (General disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 2 (2)
Implant Site Paraesthesia (General disorders) | 0 (0) | 1 (1)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 7 (7) | 4 (4)
Malaise (General disorders) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 4 (5) | 2 (2)
Pain (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Sensation Of Foreign Body (General disorders) | 1 (1) | 1 (1)
Sensation Of Pressure (General disorders) | 1 (1) | 0 (0)
Spinal Pain (General disorders) | 0 (0) | 2 (2)
Swelling (General disorders) | 1 (1) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Latex Allergy (Immune system disorders) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Adenoviral Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 3 (4)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia Primary Atypical (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1)
Reiter's Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 5 (5)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 1 (1)
Stitch Abscess (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (2) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dural Tear (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Electric Shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (10) | 27 (28)
Foreign Body (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Graft Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Erythema (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Oedema (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incorrect Dose Administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intervertebral Disc Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Nail Avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Constipation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypertension (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Road Traffic Accident (Injury, poisoning and procedural complications) | 7 (7) | 15 (15)
Spondylopathy Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal Deviation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound Contamination (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Secretion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Blood Cholesterol Increased (Investigations) | 2 (2) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 3 (3)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Blood Triglycerides Increased (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T Wave Abnormal (Investigations) | 1 (1) | 0 (0)
Haematocrit Decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Intraocular Pressure Test Abnormal (Investigations) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 (0) | 1 (1)
Reflex Test Abnormal (Investigations) | 0 (0) | 1 (1)
Sleep Study Abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Urine Output Decreased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gout (Investigations) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 14 (14)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 29 (34) | 44 (47)
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (13)
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 12 (15) | 20 (21)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 18 (21) | 26 (27)
Intervertebral Disc Space Narrowing (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint Crepitation (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Joint Hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Laxity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 21 (24) | 40 (46)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 4 (5) | 11 (13)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (12)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 11 (13) | 11 (12)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 37 (42) | 67 (77)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 9 (10) | 21 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 24 (27)
Myofascial Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Myofascial Spasm (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck Mass (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 63 (68) | 106 (122)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 33 (37) | 64 (72)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 29 (29)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (10)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensation Of Heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (12) | 11 (16)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibrous Cortical Defect (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous System Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Allodynia (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Arachnoid Cyst (Nervous system disorders) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1) | 1 (1)
Burning Sensation (Nervous system disorders) | 4 (4) | 7 (7)
Carpal Tunnel Syndrome (Nervous system disorders) | 10 (10) | 16 (16)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cervical Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 5 (5)
Cervicogenic Headache (Nervous system disorders) | 1 (1) | 0 (0)
Coordination Abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Cubital Tunnel Syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 7 (8)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 4 (4) | 3 (3)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 25 (26) | 39 (41)
Horner's Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hyperpathia (Nervous system disorders) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 0 (0) | 2 (2)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 34 (42) | 71 (97)
Intracranial Hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 3 (3)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 5 (5) | 6 (6)
Muscle Contractions Involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 3 (3)
Narcolepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 0 (0) | 2 (2)
Nerve Root Compression (Nervous system disorders) | 0 (0) | 2 (2)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 21 (25) | 45 (51)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Piriformis Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Post-Traumatic Headache (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radicular Pain (Nervous system disorders) | 1 (1) | 21 (21)
Radicular Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2)
Sensory Disturbance (Nervous system disorders) | 0 (0) | 2 (2)
Sensory Loss (Nervous system disorders) | 1 (1) | 5 (5)
Sinus Headache (Nervous system disorders) | 1 (1) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Tension Headache (Nervous system disorders) | 1 (1) | 1 (1)
Thoracic Outlet Syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 2 (2)
Ulnar Neuritis (Nervous system disorders) | 0 (0) | 3 (3)
Viith Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vocal Cord Paralysis (Nervous system disorders) | 1 (1) | 3 (3)
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Affect Lability (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 7 (8)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 10 (10) | 10 (10)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 7 (7)
Libido Decreased (Psychiatric disorders) | 2 (2) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 3 (3) | 2 (2)
Stress (Psychiatric disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menopausal Symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Physical Assault (Social circumstances) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Suture Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral Coldness (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less